CLINICAL TRIAL: NCT06303700
Title: Dyspnea, Risk of Falling and Quality of Life in Adolescents, Youth and Geriatric Groups
Status: Completed | Type: Observational
Sponsor: Amira Hussin Hussin Mohammed (Other)
Responsible Party: Sponsor-Investigator, Amira Hussin Hussin Mohammed, Associated professor at faculty of physical therapy, Delta University for Science and Technology
Organization: Delta University for Science and Technology (Other)
Other Study IDs: Quality of life
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Public Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- adolescents: from both sex, age ranged from twelve to seventeen years old, free from mobility disability and Severe cognitive impairment
- youth: from both sex, age ranged from twenty to twenty-two years old, free from mobility disability and Severe cognitive impairment
- geriatrics: from both sex, age ranged from sixty to eighty years old, free from mobility disability and Severe cognitive impairment

SUMMARY:
To assess the correlation between aspects of the dyspnea scale (indicating poor functionality), the fall efficacy scale (indicating a higher fear of falling), and all aspects of the SF36 (indicating quality of life) in 3 age groups: adolescents, youth, and geriatrics.

DETAILED DESCRIPTION:
An observational study was done to assess the correlation between aspects of the dyspnea scale (indicating poor functionality), the fall efficacy scale (indicating a higher fear of falling), and all aspects of the SF36 (indicating quality of life) in 3 age groups: adolescents, youth, and geriatrics. The participants in each group were assessed using the previously mentioned scales. Then the relationships between them were calculated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

The participants were male or female community-dwellers, They ranged in age: adolescents from 12 to 17 years old, youth from 20 to 22 years old, and geriatrics from 60 to 80 years old.

Exclusion Criteria:

subjects with mobility disabilities and severe cognitive impairments.

Ages: 12 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All subjects were recruited from inhabitants of urban and rural areas in the Nile Delta Region, Egypt. They were assigned into 3 age-difference groups (adolescents, youth, and geriatrics).
Sampling Method: Probability Sample
Enrollment: 604 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
the severity of dyspnea | At the baseline evaluation
  Using a dyspnea 12 (D-12) questionnaire that assesses the severity of dyspnea using a rubric of the physical and emotional aspects of dyspnea.
the level of fear of falling through daily life activities | At the baseline evaluation
  Using Fall efficacy scale (FES-I) questionnaire that assesses the level of fear of falling through daily life activities
quality of life and public health | At the baseline evaluation
  Using the Short Form 36 (SF-36) questionnaire. The questionnaire was assigned to eight domains: physical functioning, role-functioning, bodily pain, general health, vitality, social functioning, and role-emotional and mental health

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt